CLINICAL TRIAL: NCT04405674
Title: A Phase II Two Cohorts Prospective Study to Evaluate the Efficacy and Safety of Tislelizumab Combined With Chemotherapy With or Without Bevacizumab in Non-squamous NSCLC With EGFR Sensitizing Mutation Who Failed EGFR TKI Therapy
Brief Title: Tislelizumab Combined With Chemotherapy With or Without Bevacizumab in TKI-Resistant EGFR-Mutated Non-squamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Professor, Director of Pulmonary Medicine at Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2001-IIT
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Tislelizumab; PD-1; Chemotherapy; EGFR mutation; Non small cell lung cancer; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Carboplatin; Pemetrexed; Bevacizumab; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tislelizumab plus chemotherapy (Experimental): Tislelizumab plus Carboplatin/Nab-paclitaxel as induction treatment and followed by Tislelizumab plus pemetrexed as maintenance treatment.
  Interventions: Drug: Tislelizumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Nab paclitaxel
- Tislelizumab plus chemotherapy plus Bevacizumab (Experimental): Tislelizumab plus Nab-paclitaxel and Bevacizumab as induction treatment and followed by Tislelizumab plus Bevacizumab as maintenance treatment.
  Interventions: Drug: Tislelizumab; Drug: Bevacizumab; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: BGB-A317
Drug: Carboplatin — Carboplatin AUC 5 administered intravenously (IV) on Day 1 of each 21-day cycle, 4 cycles
  Arms: Tislelizumab plus chemotherapy
Drug: Pemetrexed — Pemetrexed 500mg/m2 administered intravenously (IV) on Day 1 of each 21-day cycle
  Arms: Tislelizumab plus chemotherapy
Drug: Bevacizumab — Bevacizumab 7.5mg/kg administered intravenously (IV) on Day 1 of each 21-day cycle
  Arms: Tislelizumab plus chemotherapy plus Bevacizumab
Drug: Nab paclitaxel — Nab-paclitaxel 260mg/m2 administered intravenously (IV) on Day 1 of each 21-day cycle, 4 cycles

SUMMARY:
A phase II, open-label, multicenter, two cohorts, prospective clinical study to investigate the efficacy and safety of tislelizumab (anti-pd1 antibody) combined with chemotherapy with or without bevacizumab in non-squamous non-small cell lung cancer patients with EGFR sensitizing mutation who failed EGFR TKI (Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor) therapy.

DETAILED DESCRIPTION:
Although EGFR tyrosine kinase inhibitors (TKI) have improved the survival of EGFR mutated NSCLC pts, drug resistance inevitably develops in almost all pts. Tislelizumab (tis), an anti-PD-1 mAb, has shown improved efficacy when combined with chemotherapy in pts with advanced EGFR-wt NSCLC with a tolerable safety profile. This study aims to evaluate the efficacy and safety of tislelizumab plus carboplatin and Nab-paclitaxel（cohort 1）or tislelizumab plus Nab-paclitaxel and bevacizumab （cohort 2） in EGFR-mut nsq-NSCLC pts failed to EGFR TKI therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, locally advanced (Stage IIIB/C) not amenable to curative surgery or radiotherapy, or metastatic (Stage IV) non-squamous NSCLC according to American Joint Committee on Cancer, 8th Edition.
2. Documentation of tumor EGFR sensitizing mutation before EGFR TKI treatment, including 19del, L858R, G719X, S786I and L861Q.
3. Disease progression after treatment with an EGFR TKI therapy: 1) Patients previously treated with 1st or 2nd generation EGFR TKI (e.g. erlotinib/afatinib/gefitinib/icotinib) are required to provide specimens after PD to confirmed absence of EGFR T790M mutation; 2) Patients with confirmed acquired T790M mutation after 1st or 2nd generation EGFR TKI (e.g. erlotinib/afatinib/gefitinib/icotinib) are required to have 3rd generation EGFR TKI (e.g. osimertinib) treatment failure prior to enrollment; 3) Patients previously failed from 3rd generation EGFR TKI (e.g. osimertinib) treatment as 1st line therapy are eligible regardless of their EGFR T790M mutation status.
4. ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1.
5. Life expectancy ≥ 3 months.
6. Adequate organ function
7. Able to provide written informed consent by the patient or by the patient's legally acceptable representative and can understand and agree to comply with the requirements of the study.
8. 18 to 75 years old on the day of signing the ICF (Informed Consent Form).

Exclusion Criteria:

1. Received prior therapies targeting PD-1, PD-L1, CTLA-4 or other immune checkpoints.
2. Received prior platinum-based chemotherapy for advanced disease.
3. Patients who have received prior systemic anti-vascular therapy (e.g., bevacizumab and small molecule VEGFR inhibitors) for advanced disease (Cohort 2)
4. Received EGFR TKI treatment within 2 weeks
5. Treatment with any approved systemic anti-cancer therapy or systemic immune-stimulatory agents (including but not limited to interferons, interleukin IL-2, and tumor necrosis factor) within 28 days prior to initiation of study treatment.
6. Clinically uncontrolled pleural effusion or ascites that requires pleurocentesis or abdominal tapping for drainage within 2 weeks prior to initiation of study treatment.
7. Active leptomeningeal disease or uncontrolled brain metastasis.
8. History of allergic reactions to any study drugs.
9. CrCl < 45 mL/min
10. Patients with active viral hepatitis that requires treatment.
11. Active autoimmune diseases that requires treatment and may affect study treatment estimated by investigator.
12. Any condition that required systemic treatment with either corticosteroids or any other immunosuppressive medication that may affect study treatment estimated by investigator.
13. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy.
14. History of hemoptysis, i.e., coughing up at least one-half teaspoon of fresh blood, within 3 months prior to enrollment. (Cohort 2)
15. Imaging shows tumor invasion of a large vessel (e.g., pulmonary artery or superior vena cava) that the investigator determines is at risk for bleeding. (Cohort 2)
16. Had minor surgical procedures, such as tube placement, within 48 hours prior to first bevacizumab treatment. (Cohort 2)
17. Recently treated with a full dose oral or parenteral anticoagulant or thrombolytic agent. Prophylactic using anticoagulants is allowed. (Cohort 2)
18. History or test results indicating an inherited bleeding tendency or coagulation disorder that may increase the risk of bleeding (cohort 2)
19. uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) (cohort 2)
20. Clinically meaningful (e.g., active) cardiovascular disease that, in the judgment of the investigator, is intolerant to bevacizumab therapy (cohort 2)
21. Non-cured wound, peptic ulcer in active phase, or fracture (cohort 2)
22. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or thrombotic disease within 6 months judged by the investigator to be intolerant to bevacizumab treatment (Cohort 2)
23. With a history of interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung diseases, etc.
24. Have known human immunodeficiency virus (HIV) infection.
25. Any major surgical procedure requiring general anesthesia ≤ 28 days before initiation of study treatment.
26. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that would be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs (Adverse Events) or result in insufficient or might impair compliance with study conduct.
27. Concurrent participation in another clinical study.
28. Pregnant or lactating women, or male and female patients who plan to have children during the study period. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
1-Year Progression-Free Survival Rate (1-Year PFS Rate) | up to 24 months after enrollment or study close
  Progression-free survival (per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first. Subjects who do not have disease progression will be censored at their last valid tumor assessment. PFS rate at 1 year as estimated by Kaplan-Meier method.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 24 months after enrollment or study close
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first.
Objective Respond Rate (ORR) | up to 24 months after enrollment or study close
  ORR (per RECIST 1.1) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | up to 24 months after enrollment or study close
  DCR (per RECIST 1.1) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD).
Overall Survival (OS) | up to 24 months after enrollment or study close
  OS is defined as the time from the starting date of study drug to the date of death due to any cause.
Duration of Response (DoR) | up to 24 months after enrollment or study close
  DoR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China